CLINICAL TRIAL: NCT01321346
Title: A Phase I Dose Finding Study Of Panobinostat In Children With Refractory Hematologic Malignancies
Brief Title: A Study Of Panobinostat In Children With Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2009-012
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood; Myelogenous Leukemia, Acute, Childhood; Hodgkin's Disease; Non-Hodgkin's Lymphoma
Keywords: Relapse; Lymphoblastic; Leukemia; Panobinostat; LBH589; Refractory; Hodgkin's; Non-Hodgkin's Lymphoma; Lymphoma; Myelogenous; Acute; Childhood; Pediatric; ALL; AML; NHL; HD
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid; Hodgkin Disease; Lymphoma, Non-Hodgkin; Recurrence; Leukemia; Lymphoma | interventions — Panobinostat; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Leukemia Patients (Experimental): Patients with ALL and AML will be treated in one arm of the study.
  Interventions: Drug: Panobinostat; Drug: Cytarabine
- Lymphoma Patients (Experimental): Patients with NHL or HD will be treated in one arm of the study.
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Dose will be assigned at study entry. Patients will take panobinostat orally 3 times a week given on a Monday, Wednesday, Friday schedule, every week. One course is 28 days (4 weeks). Patients will get 2 courses and may receive up to 8 courses total.
  Other Names: LBH589
  Arms: Leukemia Patients
Drug: Cytarabine — All patients will receive 70 mg of intrathecal cytarabine on day "0" of course 1. The day "0" dose must be given at least 24 hours prior to initiation of panobinostat. Omit the day "0" dose of intrathecal cytarabine if the patient received intrathecal therapy within 72 hours of treatment.
  All patients will receive 70 mg of intrathecal cytarabine on day "29" of course 1-8 in conjunction with their disease evaluation.
  Other Names: Ara-C; cytosine arabinoside; Cytosar
  Arms: Leukemia Patients
Drug: Panobinostat — Dose will be assigned at study entry. Patients will take panobinostat orally 3 times a week on a Monday, Wednesday, Friday schedule, every other week. Once course is 28 days (4 weeks). Patients will get 2 course and may receive up to 8 courses of therapy.
  Other Names: LBH589
  Arms: Lymphoma Patients

SUMMARY:
This study is for patients with relapsed or refractory Acute Lymphoblastic Leukemia (ALL), Acute Myelogenous Leukemia (AML), Hodgkin's Disease (HD) or Non-Hodgkin's Lymphoma (NHL). Panobinostat is a new drug that is considered investigational because it has not been approved in the United States by the Food and Drug Administration (FDA), or in any other country. Panobinostat is a histone deacetylase inhibitor (HDACi) and interferes with gene expression found in cells causing them to stop growing or die. Panobinostat has been used in several hundred adults who had leukemia, HD, NHL and other solid tumors. Panobinostat has not been given to children.

This is a phase I study. In a phase I study, drugs are tested to the highest dose that can be safely given. Drugs are given at gradually increasing dosages until there are unacceptable side effects. The goal of the Phase I study is to find out the dose of panobinostat that can be safely given to children with relapsed ALL, AML, HD and NHL.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≤ 21 years of age at the time of enrollment.
* Patients must have one of the following:

  1. Patient must have relapsed/refractory acute myelogenous leukemia (AML) with ≥ 5% blast in the bone marrow or biopsy confirmed chloroma. Patient may have CNS 1, 2 or 3 disease. Isolated CNS relapse is not eligible.
  2. Patient must have relapsed/refractory acute lymphoblastic leukemia (ALL) with ≥ 5 blasts in the bone marrow or biopsy confirmed extramedullary disease. Patient may have CNS 1, 2 or 3 disease. Isolated CNS relapse is not eligible.
  3. Patient must have relapsed or refractory non-Hodgkin's lymphoma (NHL) or Hodgkin's disease. Patients must have CNS 1 disease. Patient must have histologic verification of disease at original diagnosis. Patient must have measurable disease documented by clinical or radiographic criteria or bone marrow disease present at study entry.
* Karnofsky > 50% for patients > 16 years of age and Lansky > 50% for patients less than or equal to 16 years of age. (See Appendix I for Performance Scales).
* Patient must have a life expectancy of 8 weeks.
* PRIOR THERAPY Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  1. Patients with AML must have had at least 2 prior therapeutic attempts including frontline induction.
  2. Patients with ALL must have had at least 3 prior therapeutic attempts including frontline induction.
  3. Radiotherapy: At least 28 days must have elapsed since and radiation therapy.
  4. Hematopoietic Stem Cell Transplant:

     Patients who have had previous allogeneic HSCT must have grade I or less of Graft-versus-Host Disease (GVHD) and have not received immunosuppressive medication for at least 90 days.
  5. Hematopoietic grow factors: It must have been at least 7 days since the completion of therapy with GCSF or other growth factors at the time of enrollment. It must have been at least 14 days since the completion of therapy with pegfilgrastim (Neulasta®).
  6. Biologic/Immunologic (anti-neoplastic) therapy: It must be at least 28 days since the completion of therapy with a biologic/immunologic agent such as a monoclonal antibody prior to study enrollment and at least 28 days since non-study chemotherapy has been administered, excluding CNS directed therapy as described in Section 4.1.
  7. Prior HSCT for Hodgkin's Lymphoma: Patients with Hodgkin's lymphoma must have had prior attempt at autologous HSCT.
* Renal and Hepatic Function

  1. Patient's serum creatinine must be ≤ 1.5 x institutional upper limit of normal (ULN) according to age. If the serum creatinine is greater than 1.5 times normal, the patient must have a calculated creatinine clearance or radioisotope GRF ≥ 70mL/min/1.73m2.

     * Pediatric Population (age <18): Calculated creatinine clearance ≥ 90 ml/min/1.73m2 as calculated by the Schwartz formula for estimated glomerular filtration rate (GFR)
     * Adult Population (age >18): Serum creatinine <1.0 mg/dL; if serum creatinine >1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be >60 mL/min/1.73 m2
  2. Patient's ALT must be < 5 x institutional upper limit of norm ULN.
  3. Patient's total bilirubin must be ≤ 1.5 x ULN.
* Cardiac Function

  a. Patient must have a shortening fraction ≥ 29% or an ejection fraction ≥ 40% by ECHO/MUGA.
* Reproductive Function

  1. Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
  2. Female patients with infants must agree not to breastfeed their infants while on this study.
  3. Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study.

Exclusion Criteria:

* Patients will be excluded if they are unable to swallow capsules whole.
* Patients will be excluded if they have received previous therapy with HDAC, DAC, HSP90 inhibitors or valproic acid anticancer therapy. Valproic acid therapy is not allowed for any reason while on this study.
* AML patients who are candidates for allogeneic stem cell transplant are excluded.
* Patients will be excluded if they have a systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment.
* Gastrointestinal Function

  1. Impairment of GI function or GI disease that may significantly alter the absorption of panobinostat.
  2. Patients with diarrhea > CTCAE grade 2.
* Patients will be excluded if there is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period, excluding CNS directed therapy upfront for AML patients and continuing for CNS positive patients as described in Section 4.1. Cyto-reduction with hydroxyurea can be initiated and continued for up to 24 hours prior to the start or protocol therapy.
* Patients will be excluded if they have significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required.
* Cardiac Exclusion Criteria:

Patients will be excluded if these meet any of the following:

1. History or presence of sustained ventricular tachyarrhythmia. (Patients with a history of atrial arrhythmia are eligible but should be discussed with the study chair prior to enrollment).
2. Any history of ventricular fibrillation or torsade de pointes.
3. Bradycardia defined as HR< 50 bpm. Patients with pacemakers are eligible if HR ≥ 50 bpm.
4. Screening ECG with a QTc > 450 msec.
5. Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug.
6. Right bundle branch block + left anterior hemiblock (bifascicular block).
7. Patients with myocardial infarction or unstable angina ≤ 6 months prior to starting study drug.
8. Other clinically significant heart disease (e.g., CHF NY Heart Association class III or IV, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen).
9. Patients with leukemia must not be known to be refractory to red blood cell or platelet transfusions.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
To find the highest dose of oral panobinostat that can be given to patients with relapsed AML, HD or NHL without causing severe side effects. | 8 weeks
To learn what kind of side effects panobinostat can cause when taken by children with relapsed ALL, AML, HD or NHL. | 8 weeks

SECONDARY OUTCOMES:
To determine whether panobinostat is a beneficial treatment for ALL, AML, HD or NHL. | 8 weeks
To test the amount of panobinostat in the patient's blood and spinal fluid after taking panobinostat. | 3 years
To test samples of cancer cells to see if they have chemicals that affect the way panobinostat works. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Julio Barredo, MD, Study Chair — University of Miami
Locations (20):
- United States (20):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - UCSF School of Medicine, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami Cancer Center, Miami, Florida
  - Children's Healthcare of Atlanta, Emory University, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Dana Farber, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Childrens Hospital & Clinics of Minnesota, Minneapolis, Minnesota
  - New York University Medical Center, New York, New York
  - Children's Hospital New York-Presbyterian, New York, New York
  - Levine Children's Hospital at Carolinas Medical Center, Charlotte, North Carolina
  - Rainbow Babies, Cleveland, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - St. Jude, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Primary Children's, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Goldberg J, Sulis ML, Bender J, Jeha S, Gardner R, Pollard J, Aquino V, Laetsch T, Winick N, Fu C, Marcus L, Sun W, Verma A, Burke M, Ho P, Manley T, Mody R, Tcheng W, Thomson B, Park J, Sposto R, Messinger Y, Hijiya N, Gaynon P, Barredo J. A phase I study of panobinostat in children with relapsed and refractory hematologic malignancies. Pediatr Hematol Oncol. 2020 Sep;37(6):465-474. doi: 10.1080/08880018.2020.1752869. Epub 2020 Apr 27. PMID 32338562
- See also: TACL Consortium Web Site — http://tacl.us